CLINICAL TRIAL: NCT02632838
Title: Utilizing a Mobile Health (mHealth) Application to Improve Hypertension Monitoring and Self-management in an Underserved Community: A Pilot Study
Brief Title: Improve Hypertension Monitoring and Self-management by Using mHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Peijia Zha, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro20150001419
Record Dates: First submitted 2015-12-03; First posted 2015-12-17 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-04

CONDITIONS: Hypertension
Keywords: Hypertension; mHealth; underserved community
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- the mHealth Group (Experimental): The mHealth group will ask to use iHealth BP7-Wireless Blood Pressure Wrist Monitor on a daily basis at HOME and also will be asked to visit community health center once a week to receive the regular hypertension care for the 6-month period as usual.
  Interventions: Device: iHealth BP7-Wireless Blood Pressure Wrist Monitor,
- the Standard Follow-up Group (No Intervention): The standard follow-up group will receive regular hypertension care as usual which consists: nursing assessment, medication management, patient education, follow up and continuing care in the community health center

INTERVENTIONS:
Device: iHealth BP7-Wireless Blood Pressure Wrist Monitor, — The mHealth group will ask to use iHealth BP7-Wireless Blood Pressure Wrist Monitor at home. This monitor is a fully automatic wrist cuff blood pressure monitor that uses the oscillometric principle to measure blood pressure and pulse rate. The monitor works with mobile devices to test, track and share vital blood pressure data. The Bluetooth sync system allows the monitor to send BP measures and pulse rate to patients' mobile devices. The free iHealth app automatically keeps a history of BP data and gives patient the option to share their blood pressure data with their provider. In addition to keep the data on the mobile device, patient also receive a free and secure cloud account. Vital data on the cloud allows patients to access from any computer and to share with their provider.
  Other Names: 510(k) number: 121470
  Arms: the mHealth Group

SUMMARY:
Monitoring and self-management are important components of effective chronic disease care and improved patient outcomes. With the rapid development of integration of mobile health technology (mHealth) into health care delivery services, mHealth intervention provides a great opportunity to improve the efficiency of chronic disease management. However, little is known about whether mHealth interventions can effectively impact the health and health care outcomes in underserved populations. This pilot study will assess the preliminary effectiveness of a mobile-based health intervention in an urban underserved community with a high incidence of hypertension. It is hypothesized that patients with hypertension will experience improved outcomes due to the use of a mHealth application compared with patients who are not using the application. The findings from this study will advance our understanding of the utility of mHealth interventions among underserved populations and generate evidence to support this new health care delivery approach in underserved urban communities.

In this study, two hypotheses will be tested:

1. Hypertension patients using the mHealth application exhibit a greater decrease in blood pressure and better maintenance over a 6-month period compared to those who receive standard care.
2. Hypertension patients using the mHealth application will exhibit more effective self-management as compared to those who receive standard care.

DETAILED DESCRIPTION:
Based on the J&HCHC's current practice, all hypotension patients are required to visit the nurses for their regular hypertension care every week. Therefore, all participants in this study will be asked to visit J&HCHC once a week for the 6-month period as usual. The standard follow-up group will receive regular hypertension care as usual which consists: nursing assessment, medication management, patient education, follow up and continuing care. Home monitoring is a great way to help detect and monitor high blood pressure. The mHealth group will ask to use iHealth BP7-Wireless Blood Pressure Wrist Monitor on a daily basis at HOME and also will be asked to visit J&HCHC once a week to receive the regular hypertension care for the 6-month period as usual. After all participants complete their 6-month study, the study data will be collected from Electronic Health Record (McKesson) and patient's mobile devices.

In this study, a FDA 510K approved device, iHealth BP7-Wireless Blood Pressure Wrist Monitor (iHealth Lab Inc.), will be utilized for the mHealth group. This is a fully automatic wrist cuff blood pressure monitor that uses the oscillometric principle to measure blood pressure and pulse rate. The monitor works with mobile devices to test, track and share vital blood pressure data. There are no physical risks associated with using this device to take the blood pressure at home. Besides the FDA 510K approval, iHealth BP7-Wireless Blood Pressure Wrist Monitor has also CE medical certification (Europe) and ESH Certification (European Society of Hypertension). iHealth BP7-Wireless Blood Pressure Wrist Monitor works with both Apple and Android devices. Apple iOS devices requires iOS version 5.0 or higher and Android devices requires operating system 3.0 or later.

iHealth BP7-Wireless Blood Pressure Wrist Monitor can maintain a maximum of 10,000 measurements or three years of usage. In addition, iHealth BP7-Wireless Blood Pressure Wrist Monitor has a Bluetooth sync system that will pair with both Apple and Android devices. The synchronization allows the monitor to send systolic and diastolic blood pressures and pulse rate to patients' mobile devices. The free iHealth MyVitals app then automatically keeps a history of BP data and gives patient the option to share their blood pressure data information with their healthcare provider. In addition to keep the data on the mobile device, patient also receive a free and secure cloud account. Vital data on the cloud allows patients to access from any computer and to share readings with their healthcare provider, if they choose to do so. With this type of information available, patients will be able to do self-management and nurses will be able to actively provide intervention activities. Conceptual diagram for iHealth BP-7 Wireless Blood Pressure Wrist Monitor device, apps and cloud sever are presented in research protocol

A pilot version of a parallel-group 6-month randomized controlled trial (RCT) will be utilized to this study. 30 participants will be randomly assigned either to standard care and treatment (the standard follow up group) or to the mobile intervention group (the mHealth group). For the standard follow up group, participants' BP will be measured in an upright seated position with feet flat on the floor while being at rest for at least 5 minutes. During each visit, participants will be measured twice or more, separated by two minutes in each arm. The Welch Allyn Spot Vital Signs LXi electronic blood pressure monitor will be utilized for this group. Participants' systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse will be measured and recorded by the J&HCHC nurses. For the mHealth group participants' BP data will be collected in two ways: iHealth's MyVitals and office visit BP records. The office visit BP will be measured in a manner identical to the standard follow up group. iHealth's MyVitals BP data were collected by a project research assistant every week. Data were aggregated, and an average of the BP readings recorded at baseline (beginning of the study), at three months and six months will be used for data analysis.

BP monitoring adherence for the standard follow-up group will be calculated by dividing the total number of office visits to measure BP by the total number of expected visits (one office BP measurement every week for 6 months). BP monitoring adherence for the mHealth group will be calculated by dividing the total number of times iHealth BP-7 was used to measure BP by the total number of expected times it should have been used (one BP measurement performed every day for 6 months).

Improved health related quality of life, patient self-efficacy, and reduced hospital utilization will be measured. Medical Outcomes Study 36-Item Short- Form Health Survey (SF-36) will be utilized to measure the health-related quality of life. Patient self-efficacy and treatment adherence will be measured by the Medication Adherence Self-Efficacy Scale (MASES). Self-reported hospital utilization rate will be used to measure reduced hospital utilization. Participants hospital utilization data will be retrieved from their electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

1)18-64 year-old residents of one of the three housing developments and use our community health center as their primary care service

2) Subjects who have been documented with uncontrolled blood pressure, and whose BP measures 140/90 mmHg or higher for either of the two numbers

3) Subjects must have a compatible mobile device

4) Nurses in this study must be who are currently working at our community health center

Exclusion Criteria:

1. Patients under the age of 18 years old
2. Pregnant women
3. Patient with serious arrhythmia
4. Patient with preeclamptic
5. Patient who cannot speak/read English.
6. Patients using University Hospital or other clinical offices as their primary care service

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peijia Zha, PhD, Principal Investigator — Rutgers University
Locations (1):
- Peijia Zha, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited though recruitment flyers, nurses and community health workers (CHWs). Potential participants were invited to attend the information session held by the research team. Informed consent and Health Insurance Portability and Accountability Authorization were obtained for those who were eligible to participate in the study.
Pre-assignment Details: We have total 30 participants enrolled in the study, there was no significant events occurred before they were assigned to groups.
Groups:
- the mHealth Group: The mHealth group will ask to use iHealth BP7-Wireless Blood Pressure Wrist Monitor on a daily basis at HOME and also will be asked to visit community health center once a week to receive the regular hypertension care for the 6-month period as usual.
  iHealth BP7-Wireless Blood Pressure Wrist Monitor,: The mHealth group will ask to use iHealth BP7-Wireless Blood Pressure Wrist Monitor at home. This monitor is a fully automatic wrist cuff blood pressure monitor that uses the oscillometric principle to measure blood pressure and pulse rate. The monitor works with mobile devices to test, track and share vital blood pressure data. The Bluetooth sync system allows the monitor to send BP measures and pulse rate to patients' mobile devices. The free iHealth app automatically keeps a history of BP data and gives patient the option to share their blood pressure data with their provider. In addition to keep the data on the mobile device, patient also receive a free and secure cloud account. Vi
Period: Overall Study
Arm/Group | the mHealth Group | the Standard Follow-up Group
Started | 15 | 15
Completed | 12 | 13
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: 30 participants were randomly assigned in the mHealth group and the standard follow-up group. 15 in each group.
Groups:
- the mHealth Group: The mHealth group asked to use iHealth BP7-Wireless Blood Pressure Wrist Monitor on a daily basis at HOME and also asked to visit community health center once a week to receive the regular hypertension care for the 6-month period as usual.
- the Standard Follow-up Group: The standard follow-up group received regular hypertension care as usual which consists: nursing assessment, medication management, patient education, follow up and continuing care in the community health center
- Total: Total of all reporting groups
Arm/Group | the mHealth Group | the Standard Follow-up Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants] — Population: Three participants in the mHealth group withdrew the study, two participants in the standard follow-up group lost follow up. The final analysis included 25 participants.
  Participants
    number analyzed (Participants) | 12 | 13 | 25
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 12 | 13 | 25
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Three participants in the mHealth group withdrew the study, two participants in the standard follow-up group lost follow up. The final analysis included 25 participants.
  years
    number analyzed (Participants) | 12 | 13 | 25
    (all) | 48.9 (8) | 55.5 (5.2) | 52.4 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Three participants in the mHealth group withdrew the study, two participants in the standard follow-up group lost follow up. The final analysis included 25 participants.
  Participants
    number analyzed (Participants) | 12 | 13 | 25
    Female | 12 | 12 | 24
    Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Three participants in the mHealth group withdrew the study, two participants in the standard follow-up group lost follow up. The final analysis included 25 participants.
  Participants
    number analyzed (Participants) | 12 | 13 | 25
    Hispanic or Latino | 0 | 1 | 1
    Not Hispanic or Latino | 12 | 12 | 24
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Three participants in the mHealth group withdrew the study, two participants in the standard follow-up group lost follow up. The final analysis included 25 participants.
  Participants
    number analyzed (Participants) | 12 | 13 | 25
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 12 | 12 | 24
    White | 0 | 1 | 1
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: Three participants in the mHealth group withdrew the study, two participants in the standard follow-up group lost follow up. The final analysis included 25 participants.
  Participants
    United States: number analyzed (Participants) | 12 | 13 | 25
    United States | 12 | 13 | 25
Blood Pressure (BP) [Mean (Standard Deviation); unit: mm Hg] — At the baseline, all study participants' blood pressure were measured in an upright seated position with feet flat on the floor while being at rest for at least 5 minutes. Participants were measured twice or more, separated by two minutes in each arm. The Welch Allyn Spot Vital Signs LXi electronic blood pressure monitor was utilized for this group. An average of the BP readings recorded. Population: Three participants in the mHealth group withdrew the study, two participants in the standard follow-up group lost follow up. The final analysis included 25 participants.
  mm Hg
    Systolic BP_Baseline: number analyzed (Participants) | 12 | 13 | 25
    Systolic BP_Baseline | 145.77 (5.10) | 145.67 (3.68) | 145.72 (4.32)
    Diastolic BP_Baseline: number analyzed (Participants) | 12 | 13 | 25
    Diastolic BP_Baseline | 90.48 (7.58) | 90.30 (6.46) | 90.39 (7.09)
Health-Related Quality of Life [Mean (Standard Deviation); unit: units on a scale] — Health-Related Quality of Life were measured by 36-Item Short Form Health Survey (SF-36). SF-36 consisted of the sum scores of eight subscales(physical functioning, physical role limitations, mental health, emotional role limitations, social functioning, vitality, pain, general health perceptions), which are the weighted sums of the questions. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.The eight subscales were summarized into two composite scores: physical and mental quality of life. Population: Three participants in the mHealth group withdrew the study, two participants in the standard follow-up group lost follow up. The final analysis included 25 participants.
  units on a scale
    Physicalcomponent summary_Baseline: number analyzed (Participants) | 12 | 13 | 25
    Physicalcomponent summary_Baseline | 41.22 (8.91) | 40.19 (10.85) | 40.69 (9.77)
    Mental compent summary_Baseline: number analyzed (Participants) | 12 | 13 | 25
    Mental compent summary_Baseline | 42.16 (10.79) | 48.73 (10.26) | 45.58 (10.83)
Patient Self-efficacy [Mean (Standard Deviation); unit: units on a scale] — Medication Adherence Self-Efficacy Scale (MASES) were used to measure the patient self-efficacy in adhering to prescribed hypertension medications. MASES was developed to measure several aspects of self-efficacy, including adherence to prescribed medication for the management of hypertension. The MASES includes 26 items rated on a 3-point Likert scale (1= Not at all Sure, 2= Somewhat Sure, and 3= Very Sure). The range of this scale is from 26 to 78. A total mean score is calculated by averaging responses to all items. Higher scores indicate a great level of self-efficacy Population: Three participants in the mHealth group withdrew the study, two participants in the standard follow-up group lost follow up. The final analysis included 25 participants.
  units on a scale
    number analyzed (Participants) | 12 | 13 | 25
    (all) | 64.75 (10.85) | 64.85 (11.44) | 64.80 (10.92)
Hospital Admissions for Hypertension Related Illnesses [Number; unit: hosptial Admissions] — Data obtained from patients' electronic health records. Total number of hospital admissions for hypertension related illnesses were recorded. Population: Three participants in the mHealth group withdrew the study, two participants in the standard follow-up group lost follow up. The final analysis included 25 participants.
  hosptial Admissions
    number analyzed (Participants) | 12 | 13 | 25
    (all) | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure (BP) Change
Description: BP change defined as monthly average BP in both systolic and diastolic blood pressure decrease. BP decline were expected as early as 3 month of intervention and kept to decreasing over 6 month period.
  For the mHealth group: iHealth's MyVitals BP data were collected by a project research assistant every week. Data were aggregated, and an average of the BP readings recorded at baseline, 3-month and 6-month were used for data analysis.
  For the standard follow up group, participants' BP was measured in an upright seated position with feet flat on the floor while being at rest for at least 5 minutes. During each week's office visit, participants were measured twice or more, separated by two minutes in each arm. The Welch Allyn Spot Vital Signs LXi electronic blood pressure monitor was utilized for this group. Data were aggregated, and an average of the BP readings recorded at baseline, 3-month and 6-month were used for data analysis.
Time Frame: baseline, 3 monthly intervals over 6 months of follow up
Population: All study sample were analyzed.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | the mHealth Group | the Standard Follow-up Group
Number analyzed (Participants) | 12 | 13
mm Hg
  Systolic BP_Baseline | 145.77 (5.1) | 145.67 (3.68)
  Systolic BP_3-month | 140.55 (5.46) | 142.62 (5.69)
  Systolic BP_6-month | 137.38 (4.86) | 140.88 (5.01)
  Diastolic BP_Baseline | 90.84 (7.58) | 90.30 (6.46)
  Diastolic BP_3-month | 90.53 (7.62) | 88.95 (9.02)
  Diastolic BP_6-month | 88.08 (7.45) | 88.10 (9.41)

2. Secondary Outcome: Blood Pressure Monitoring Adherence
Description: BP monitoring adherence were used to measure hypertension status monitoring experiences BP monitoring adherence for the mHealth group was calculated by dividing the total number of times iHealth BP-7 was used to measure BP by the total number of expected times it should have been used (one BP measurement performed every day for 6 months).
  BP monitoring adherence for the standard follow-up group was calculated by dividing the total number of office visits to measure BP by the total number of expected visits (one office BP measurement every week for 6 months).
Time Frame: 6 months
Population: All study sample were analyzed.
Measure: Number; unit: adherence
Arm/Group | the mHealth Group | the Standard Follow-up Group
Number analyzed (Participants) | 12 | 13
adherence | 0.71 | 0.65

3. Other Pre Specified Outcome: Health-Related Quality of Life
Description: Health-Related Quality of Life were measured by 36-Item Short Form Health Survey (SF-36).
  The SF-36 consisted of the sum scores of eight subscales (physical functioning, physical role limitations, mental health, emotional role limitations, social functioning, vitality, pain, and general health perceptions), which are the weighted sums of the questions in each sections. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The eight subscales were summarized into two composite scores (physical and mental quality of life). Various studies demonstrated that the reliability of the SF-36 have exceeded 0.80 The SF-36 scores compared at baseline and 6-month later
Time Frame: baseline and 6-month
Population: All study sample data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- the mHealth Group; the Standard Follow-up Group: SF-36 scores between the baseline and 6-month later were compared between the mHealth group and the Standard follow-up group.
Arm/Group | the mHealth Group | the Standard Follow-up Group
Number analyzed (Participants) | 12 | 13
units on a scale
  Physical component summary_Baseline | 41.22 (8.91) | 40.19 (10.85)
  Physical component summary_6-month | 42.63 (11.21) | 44.25 (11.17)
  Mental component summary_Baseline | 42.16 (10.79) | 48.73 (10.26)
  Mental component summary_6-month | 43.11 (10.23) | 49.65 (11.87)

4. Other Pre Specified Outcome: Patient Self-efficacy
Description: Medication Adherence Self-Efficacy Scale (MASES) were used to measure the patient self-efficacy in adhering to prescribed hypertension medications. MASES was developed to measure several aspects of self-efficacy, including adherence to prescribed medication for the management of hypertension. The MASES includes 26 items rated on a 3-point Likert scale (1= Not at all Sure, 2= Somewhat Sure, and 3= Very Sure). The range of this scale is from 26 to 78. A total mean score is calculated by averaging responses to all items. Higher scores indicate a great level of self-efficacy The survey scores compared at baseline and 6 months.
Time Frame: baseline and 6-month
Population: All study sample were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- the mHealth Group; the Standard Follow-up Group: MASE scores between the baseline and 6 month later were compared between the mHealth group and the Standard follow-up group.
Arm/Group | the mHealth Group | the Standard Follow-up Group
Number analyzed (Participants) | 12 | 13
units on a scale
  Baseline | 64.85 (10.85) | 64.75 (11.44)
  6-month | 69.17 (7.77) | 61 (13.08)

5. Other Pre Specified Outcome: Hospital Admissions for Hypertension Related Illnesses
Description: Data obtained from patients' electronic health records. Total number of hospital admissions for hypertension related illnesses were compared at baseline and 6 months.
Time Frame: 6 months
Population: All study sample were analyzed
Measure: Number; unit: hospital admissions
Arm/Group | the mHealth Group | the Standard Follow-up Group
Number analyzed (Participants) | 12 | 13
hospital admissions | 4 | 5

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- the mHealth Group: The mHealth group asked to use iHealth BP7-Wirless Blood Pressure Wrist Monitor on a daily basis at HOME and also asked to visit community health center once a week to receive the regular hypertension care for the 6-month period as usual.
- the Standard Follow-up Group: The standard follow-up group received regular hypertension care as usual which consists nursing assessment, medication management, patient education, follow up and continuing care in the community health center.
Arm/Group | the mHealth Group | the Standard Follow-up Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13

LIMITATIONS AND CAVEATS:
1,Low SES, urban environment cased small sample size.2,medication for some comorbidities may cause blood pressure decrease. We did not consider other comorbidities among the participants in this study, the results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT02632838/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT02632838/SAP_001.pdf